CLINICAL TRIAL: NCT05952115
Title: Efficacy of Lumbar Motor Control Training in Treatment Of Patients With Cervicogenic Headache
Acronym: CGH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar Abd_El basset Ismail Marzok, principle investigator hagar Abd El basset Ismail Marzouk, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003835
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Cervicogenic Headache
Keywords: lumbar motor control; cervicogenic hedache; cervical stabilization exercises
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Intervention Model Description: lumbar motor control and cervical stabilization exercises
Who Masked: Investigator, Outcomes Assessor
Masking Description: opaque sealed envelop
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lumbar motor control exercises (Experimental): patients will receive lumbar motor control and cervical stabilization exercises three times a week for four weeks
  Interventions: Other: lumbar motor control exercises; Other: Cervical stabilization exercises
- cervical stabilization exercises (Active Comparator): the patients will receive cervical stabilization exercises three times a week for four weeks
  Interventions: Other: Cervical stabilization exercises

INTERVENTIONS:
Other: lumbar motor control exercises — the patients will receive lumbar motor control exercises in the form of three exercises (Abdominal draw in maneuver, side-bridge, and quadruped) and the level of difficulty increased each week. For all exercises, the number of repetitions stayed the same, but the difficulty increased each week, and we progressed to the advanced level of each of the three exercises.
  This training achieves co-contraction of the local/deep stabilizing muscles (Transversus abdominis and multifidus) and strengthening the global/large spinal stabilizers (erector spinae and obliques).
  Arms: lumbar motor control exercises
Other: Cervical stabilization exercises — The exercise program consisted of an axial elongation exercise, cranio-cervical flexion exercise, cervical extension exercise, and cervical-scapulothoracic strengthening exercise. The exercise program progressed based on the exercise tolerance of the patients by increasing the repetition of the exercise (10 reps to 15 reps to 20 reps). And for the resistive exercise, the participants change to an elastic band with greater resistance (progress to the next color resistance band). Exercises were performed for 20 min/session, and an exercise log recording the date and repetition of the exercises was maintained by the therapist for each participant.

SUMMARY:
this study will be conducted to investigate the effect of lumbar motor control training exercise on headache frequency, duration, intensity and neck functional disability in cervicogenic headache patients

DETAILED DESCRIPTION:
Cervicogenic Headache is a referred pain spreading from cervical structures supplied by the upper cervical spinal nerve roots (C1-C3), this referred pain that starts from the posterior aspect of the head and neck is usually found to be unilateral, and it also can spread to the frontal, temporal and orbital aspects of the head.The patient frequently reports having a terrible headache, having less neck range of motion, performing less well at work, and having trouble focusing, that may linger for hours. The convergence of primary sensory afferents from cervical nerve roots C1 to C3 with the afferents from the occiput and trigeminal nerve causes the underlying pathology. Because of this, the Suboccipital muscles particularly, which cervical roots C1 innervates to C3, are potential risk structures. Treatment options include posture correction, cervical and upper thoracic strengthening exercises, facet joint manipulation, ultrasound therapy, laser therapy, trigger release therapy, and cervical joint mobilization.famous exercise known as "Motor control exercise" attempts to improve the coordination and effectiveness of the muscles that support and govern the spine. It can also improve coordination between the deep neck flexors and superficial neck flexors and between core muscles of the lumbar region. fifty two patients will be randomly assigned to two equal groups; experimental group will receive lumbar motor control and cervical stabilization exercises and control group will receive cervical stabilization exercises only.

ELIGIBILITY:
Inclusion Criteria:

* The age of the subjects ranged from 20-40 years old, both genders.
* Patients with chronic mechanical neck pain with frequent cervicogenic headaches persisting for more than 3 months.
* Positive flexion rotation test.
* Unilateral head pain without side shift or bilateral head pain with dominant side headache associated with neck pain and aggravated by neck movement and/or sustained awkward head positioning
* Joint tenderness in at least one of the upper three cervical joints or the occipital region as detected by manual palpation.
* Intensity of headache is moderate to severe.
* Abnormal performance in CCFT < = 26 mmHg
* Body mass index range from 18 to 25 km/m2

Exclusion Criteria:

* Fracture or previous surgery on the vertebral column.
* Spinal stenosis.
* Disc prolapsed.
* TMJ dysfunction.
* Headache with autonomic involvement, dizziness, or visual disturbance.
* Congenital condition of the cervical spine.
* Neck pain of less than three months

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-07-16 (Estimated); Primary Completion 2023-10-16 (Estimated); Study Completion 2023-10-16 (Estimated)

PRIMARY OUTCOMES:
Headache frequency: | up to four weeks
  Headache frequency will measure as the number of days with headache in the last week, ranging from 0 to 7 days
Headache duration | up to four weeks
  Headache duration will measure in total hours and average number of hours headaches lasted in the past week
Headache intensity | up to four weeks
  The Visual Analog Scale will use to quantify the patient's pain level or intensity. these scale consists of line, usually 10 cm long, ranging from no pain at one end and worst pain at the other end

SECONDARY OUTCOMES:
neck disability | up to four weeks
  Arabic version of neck disability index will be used to measure neck disability. The NDI consists of 10 sections: pain intensity, personal care, lifting, reading, headache, concentration, work, driving, sleeping, and recreation. Each section is expressed by 6 different assertions in the range 0-5, with 0 indicating no disability and 5 indicating highest disability. The total score ranges from 0 to 50.0-4= No disability,5-14= Mild disability,15-24=Moderate disability, 25-34=Sever disability,35 or more=Complete disability.